CLINICAL TRIAL: NCT05211414
Title: The Effects of a Virtual Yoga Program on Patients With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Asimina Lazaridou, PhD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021P002534
Record Dates: First submitted 2021-09-21; First posted 2022-01-27 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Based Daily Excercise (Experimental): Subjects will be trained to perform 30 minutes of moderate level yoga daily, with instruction on breathing, self-awareness, and ways to modify poses to avoid pain. Subjects will be instructed in use of the email links to access the 30-minute instructive video. Subjects will attend weekly Zoom classes to learn additional postures and techniques, which will be reflected in their 30 minutes video (i.e. a new video for each week). At these weekly remote yoga classes, they will be asked about difficulties encountered and given advice about their personal home practice.
  Interventions: Behavioral: Yoga Based Daily Excercise
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Yoga Based Daily Excercise — Subjects will be trained to perform 30 minutes of moderate level yoga daily, with instruction on breathing, self-awareness, and ways to modify poses to avoid pain. Subjects will be instructed in use of the email links to access the 30-minute instructive video. Subjects will attend weekly Zoom classes to learn additional postures and techniques, which will be reflected in their 30 minutes video (i.e. a new video for each week). At these weekly remote yoga classes, they will be asked about difficulties encountered and given advice about their personal home practice.
  Arms: Yoga Based Daily Excercise

SUMMARY:
This research is being done to determine if remote yoga-based exercise can help reduce chronic pain. It will include three virtual research visits. This cohort study will include three remote research visits and an online questionnaire administration. In addition, participants will attend 8 weekly virtual yoga sessions with a daily 30-minute "homework assignment" of 30 minutes of video-guided yoga practice.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain for > 6 months' duration
* on stable doses of medication prior to entering the study and agree not to change medications or dosages (or CAM treatments) during the trial
* have an average pain score of 4/10 or greater over the previous week
* at least mild degree of sleep disturbance, defined as Pittsburgh Sleep Quality Index (PSQI) score >5
* are able to speak and understand English
* have access to a computer or tablet at home and have an email address
* are not currently engaged in a rigorous daily exercise routine (>5X/week)
* are willing and physically able to participate in virtual yoga-based exercise

Exclusion Criteria:

* currently under active cancer treatment (chemo, infusion, ongoing radiation)
* acute osteomyelitis or acute bone disease
* current diagnosis of chronic systemic inflammatory diseases including rheumatoid arthritis and lupus
* present or past diagnosis of schizophrenia, delusional disorder, psychotic disorder, or dissociative disorder that would be judged to interfere with study participation
* pregnancy
* any clinically unstable systemic illness judged to interfere with exercise treatment
* a pain condition requiring urgent surgery
* an active addiction disorder, such as cocaine or IV heroin use, that would interfere with study participation
* contraindications to yoga (e.g., severe back or neck injury or surgery)
* regular meditation practice or other meditative practice (e.g tai-chi, meditative form of yoga or contemplative prayer) for >20 min/week in the past 2 years
* participating in any other therapeutic trial
* other medical condition that would interfere with ability to exercise

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Feasibility | 8 weeks
  retention, attendance, yoga practice minutes
Brief Pain Inventory | 8 weeks
  Change in Pain Intensity and Interference assessed by the Brief Pain Inventory a

SECONDARY OUTCOMES:
Pain Catastrophizing | 8 weeks
  Change in pain catastrophizing as measured by the Pain Catastrophizing Scale Scored 0-52, with higher scores indicating worse outcome.
Perceived Stress | 8 weeks
  Change in perceived stress as measured by the Perceived Stress Scale Scored 0-40, with higher scores indicating worse outcome.
Mindfulness | 8 weeks
  Change in mindfulness as measured by the Five Facets of Mindfulness Questionnaire short form Scored 24-120, with higher scores indicating better outcome.
Sleep | 8 weeks
  PROMIS scale
Anxiety | 8 weeks
  Change in Anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Chesnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided